CLINICAL TRIAL: NCT06469840
Title: French Translation/Adaptation of Affordances in the Home Environnent for Motor Development Self-Report (AHEMD-SR)
Brief Title: French Translation/Adaptation of AHEMD-SR (FR-AHEMD)
Acronym: FR-AHEMD
Status: Recruiting | Type: Observational
Sponsor: Fondation Ildys (Other)
Responsible Party: Sponsor
Other Study IDs: RI2023_007
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Motor Disorders
Keywords: AHEMD-SR; Motor Development; Pediatric rehabilitation
MeSH Terms: conditions — Motor Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents: Parents of a child aged 18 to 42 months with a diagnosis of delayed motor development
- Expert group: Pediatric rehabilitation professionals

SUMMARY:
The aim of this study is to develop a French translation and adaptation of the original English version of the AHEMD-SR.

DETAILED DESCRIPTION:
The AHEMD-SR was developed in 2005 to assess the opportunities offered to children aged 18 to 42 months to support their motor development in the home environment. The questionnaire is reliable and valid and is regularly used by researchers and practitioners to assess and develop strategies to improve the stimulating properties of the home. To date, the AHEMD-SR has been translated into eight languages, but no French translation exists.

The study will include a translation of the AHEMD-SR into French and a cultural validation of the French version of the questionnaire with a sample of parents of children diagnosed with delayed motor development and a panel of paediatric rehabilitation experts.

ELIGIBILITY:
Parents Group :

Inclusion Criteria:

* Parents of a child aged 18 to 42 months with a diagnosis of delayed motor development
* Taken in charge in one of the participating centers for an intensive motor rehabilitation training
* Francophone by birth

Exclusion Criteria:

* Parent opposing participation in the study

Experts Group :

Inclusion Criteria:

* Professional
* Holding a French state diploma in the field of rehabilitation
* Participating in an intensive motor rehabilitation training in one of the participating centres.
* Proof of experience in paediatric rehabilitation (lasting 5 years).
* Francophone by birth

Non-inclusion criteria :

- Expert opposing participation in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Parents of a child aged 18 to 42 months with a diagnosis of delayed motor development
  * Pediatric rehabilitation professionals
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Reliability of the French version of the original English version of the AHEMD-SR | July 2024 - October 2024

CONTACTS AND LOCATIONS:
Overall Officials: Rodolphe BAILLY, PhD, Principal Investigator — Fondation Ildys
Locations (2):
- France (2):
  - Les Capucins Angers, Angers
  - Fondation ILDYS, Brest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sousa VD, Rojjanasrirat W. Translation, adaptation and validation of instruments or scales for use in cross-cultural health care research: a clear and user-friendly guideline. J Eval Clin Pract. 2011 Apr;17(2):268-74. doi: 10.1111/j.1365-2753.2010.01434.x. Epub 2010 Sep 28. PMID 20874835
- [Background] Rodrigues LP, Saraiva L, Gabbard C. Development and construct validation of an inventory for assessing the home environment for motor development. Res Q Exerc Sport. 2005 Jun;76(2):140-8. doi: 10.1080/02701367.2005.10599276. PMID 16128482